CLINICAL TRIAL: NCT02141464
Title: Energy Balance and Weight Gain With Ivacaftor Treatment of CFTR Gating Mutations
Brief Title: Energy Balance and Weight Gain With Ivacaftor Treatment
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-010622
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine, stool
Oversight: Data Monitoring Committee: No

SUMMARY:
Ivacaftor is a novel, FDA approved new therapy that addresses Cystic fibrosis transmembrane conductance regulator (CFTR) dysfunctions in subjects with Cystic fibrosis (CF) and "gating mutations".

The primary aim is to determine the mechanism(s) for weight gain in participants whom Ivacaftor treatment was initiated based on clinical indications by CF Care Team. This longitudinal study will assess in detail energy expenditure, weight gain, body composition, and lung function in 24 subjects ≥6 years old with CF with a gating mutation before treatment and after three months treatment with Ivacaftor. All subjects will be seen at the Children's Hospital of Philadelphia's Clinical Translational Research Center.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disease caused by mutations in the gene encoding the CF transmembrane conductance regulator (CFTR), a chloride channel. Most CF mutations either reduce the number of CFTR channels at the cell surface (synthesis or processing mutations) or impair channel function (gating or conductance mutations). Ivacaftor (Kalydeco, VX-770) is a novel, FDA approved new therapy that addresses CFTR dysfunctions in subjects with CF and "gating mutations", specifically; it potentiates CFTR channel function. For mutations like G551D that permit CFTR expression at the cell membrane but compromise its activity, Ivacaftor increases the probability that the channel is open and active. In previous randomized, double-blind, placebo controlled trials, Ivacaftor treatment resulted in clinically significantly improvements in pulmonary function, weight and body mass index (BMI), and significant decreases in sweat chloride reflective of increased CFTR activity. The improvements in lung function and weight occurred over the first 8 weeks of treatment, plateaued and were sustained over the 48 weeks of the trial. The mechanism for the rapid and sustained weight gain is not known. Several mechanisms are considered in this proposal which may result in improved energy balance and energy utilization, and weight gain. These include decreased resting energy expenditure, increased energy and fat absorption from the gut, improved pancreatic enzyme and pH secretion, and increased energy intake. Improvements in weight and BMI status are expected to result from this improvement in energy balance and utilization, with potential beneficial effects on muscle mass and function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis with one or two CFTR gating mutations
* Age: 6 years and older
* A clinical decision has been made for the subject to start Ivacaftor treatment
* In usual state of good health
* Family and subject commitment to the 3-month study protocol with two, 3-4 day visits to CHOP

Exclusion Criteria:

* FEV1 < 40% predicted
* Use of any inhibitors or inducers of cytochrome P450 (CYP) 3A
* Pregnancy or breast feeding
* Other illness affecting growth or nutritional status
* Subjects receiving total parenteral nutrition

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 24 subjects ≥6 years old with CF with a gating mutation before treatment (baseline) and after three months treatment with Ivacaftor.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Reduction in resting energy expenditure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Stallings VA, Sainath N, Oberle M, Bertolaso C, Schall JI. Energy Balance and Mechanisms of Weight Gain with Ivacaftor Treatment of Cystic Fibrosis Gating Mutations. J Pediatr. 2018 Oct;201:229-237.e4. doi: 10.1016/j.jpeds.2018.05.018. Epub 2018 Jul 18. PMID 30029855
- [Derived] Sainath NN, Schall J, Bertolaso C, McAnlis C, Stallings VA. Italian and North American dietary intake after ivacaftor treatment for Cystic Fibrosis Gating Mutations. J Cyst Fibros. 2019 Jan;18(1):135-143. doi: 10.1016/j.jcf.2018.06.004. Epub 2018 Jul 6. PMID 29983355